CLINICAL TRIAL: NCT05441917
Title: Analysis Phototherapy and Radiofrecuency Added to a Physical Therapy Program for Treatment of Cellulite
Brief Title: Phototherapy and Radiofrecuency for Cellulite
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Dissolution of the research team
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Principal Investigator, Hernán Andrés de la Barra Ortiz, Professor, Quiropraxia y Equilibrio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11062022
Record Dates: First submitted 2022-06-11; First posted 2022-07-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cellulite
Keywords: Cellulite; Carboxytherapy; Phototherapy; Radiofrequency; Manual Therapy.
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sanae with LED (Experimental): Phototherapy is related to light emission as a form of treatment for tissue and skin conditions. Its action depends on the absorption of light by chromophores, organelles present in the dermis and epidermis that give rise to cellular responses according to the different chemical reactions caused by light. The term "LED" means light emitted by a diode, thus, when the diode is subjected to an electrical current, light emission occurs (photon). Its applicability occurs in various disorders such as acne, alopecia, localized adiposity, stretch marks, cellulite, pre and postoperative, dark circles, etc. And they can also enhance treatments by promoting drainage, hydration, whitening, and rejuvenation, among other benefits.
  Interventions: Device: Sanae method with LED
- Sanae with Radiofrecuency (Placebo Comparator): Radiofrequency (RF) is considered a non-invasive therapy that enables thermal modification in the connective tissue of the skin, through dermal heating and vasodilation. Upon reaching the tissue, the current encounters resistance, and heat is produced by converting it into thermal energy. In this way, the deep dermis undergoes controlled volumetric heating, while the epidermis is preserved through cooling systems.
  Thermal damage triggers an inflammatory cascade and stimulates neocollagenesis, causing the dermis to thicken. Vasodilation, on the other hand, leads to hyperemia and lymphatic drainage in the fat tissue. The expected physiological effects are increased circulatory and nutrient supply, improving tissue hydration and oxygenation, greater metabolic and enzymatic activity, accelerating the elimination of catabolites, lipolysis, and the contraction of connective tissue.
  Interventions: Device: Sanae method with Radiofrecuency

INTERVENTIONS:
Device: Sanae method with LED — Sanae method (combination of therapies): Manual therapy, Carboxytherapy, and phototherapy.
  Arms: Sanae with LED
Device: Sanae method with Radiofrecuency — Sanae method (combination of therapies): Manual therapy, Carboxytherapy, and radiofrequency.
  Arms: Sanae with Radiofrecuency

SUMMARY:
Cellulite is a condition that consists of an edematous infiltration of connective tissue. It has multiple factors in its etiology, making it difficult to choose just one type of treatment. Thus, aiming at greater therapeutic efficiency, the association of therapies is studied. This research aims to evaluate the Sanae method for the treatment of cellulite. The sample will feature 60 participants who have different degrees of cellulite. Initially, a pilot study will be carried out with 12 patients, divided into two groups: G1-P: 6 volunteers with grade 3 cellulite and G2-P: 6 volunteers with grade 2 cellulite. At the end of this step, the sample for the new step will include 48 people from female, who also have the same characteristics as the previous groups. Again they will be divided equally into two groups: G1: 24 volunteers with grade 3 cellulite and G2: 24 volunteers with grade 2 cellulite. Assessment protocols, photographs, ultrasound, magnetic resonance imaging and questionnaires will be used. The treatment will take place 3 times a week for 50 minutes, and will consist of a combination of therapies such as Carboxitherapy using equipment from the Ibramed™ brand, model Aires™, phototherapy from the Ibramed™ brand, model Antares™, radiofrequency from the Ibramed® brand, the Neartek™ model and manual therapy, in addition, the volunteers will wear compressive shorts during treatment. A total of 15 sessions will be carried out and the reassessment will be carried out after the last session, with the repetition of all the exams mentioned and photos for analysis of the results.

DETAILED DESCRIPTION:
1. INTRODUCTION

   Cellulite affects about 85 to 98% of women of all races after the onset of puberty, suggesting a hormonal component in its pathogenesis. It is a condition that consists of an edematous infiltration of the connective tissue, followed by polymerization of the fundamental substance which, infiltrating into the fabrics, produces a consecutive fibrotic reaction. Then, cellulite occurs as a consequence of connective tissue edema and ground substance hyperpolymerization. Thus, it manifests itself in the form of nodules or plaques of varied extension and location, and may even present pain in the affected areas.

   The occurrence of multiple factors in its etiology makes it difficult to choose only one type of therapy for its treatment. Thus, aiming at greater therapeutic efficiency, the association of therapies is studied. One of the methods that can be chosen is radiofrequency, whose main mechanisms of action are dermal heating and vasodilation. The thermal action triggers an inflammatory cascade and stimulates neocollagenesis, causing the dermis to thicken. Vasodilation, on the other hand, leads to hyperemia and lymphatic drainage in the fat tissue. The association of these mechanisms improves the appearance of the skin, bringing good results to aesthetic problems.

   Another technology that can be applied in the treatment of cellulite is the use of phototherapy. Light Emitting Diodes (LEDs) are devices made up of solid semiconductors linked together and that generate light. They provide a reliable, high-power light source in narrow bands that evenly illuminate a surface. LED does not use ablative or thermal mechanism, but there is a photochemical effect, in which light is absorbed and exerts a chemical change, showing the ability to induce photobiological processes in cells. In addition, LEDs have the ability to combine wavelengths with an array of various sizes, thus stimulating a wider range of tissue types.

   In addition to these technologies, manual lymphatic drainage is a standard therapeutic tool that has been extensively studied over the years, which uses massage with gentle compressions to stimulate the removal of excess lymph that may be present in cellulite. Linked to its application, the therapist can also choose to use compression of the treated region, playing an important role in additional

   reduction, increasing the continuous pumping mechanism. Several studies prove the effectiveness of the therapies mentioned above in the treatment of EGF. However, its cause is multifactorial and it is not possible to isolate each of these factors, which together, contribute to the onset of the disorder, requiring the combination of different treatments to achieve maximum results. Thus, the purpose of this study will be to evaluate the Sanae Method for the treatment of cellulite, using a combination of therapies.
2. OBJECTIVES

   Main objective:

   ● Evaluate the Sanae method for the treatment of Cellulite.

   Specific objectives:
   * Investigate whether there is an improvement in the appearance of the region affected by cellulite through photographic and term photographic images;
   * Analyze whether there are clinical changes through PAFEG after using the Sanae method (combination of therapies);
   * Check for possible changes in skin architecture through ultrasound and magnetic resonance imaging after using the Sanae method (combination of therapies);
   * Check changes in the quality of life of patients with cellulite.
   * Check the degree of "satisfaction of the treated individual" with the results of treatment with the Sanae method.
3. JUSTIFICATION

   The scientific production has the objective of appropriating reality to better analyze it and, later, producing transformations regarding the discussion on the use of protocols with combined therapies to maximize the therapeutic effect in the treatment of cellulite. In addition to being a very relevant practical aspect, it is of importance for the academic environment, taking into account the changes caused by the pathophysiology of cellulite, in addition to its great impact on society.

   Cellulitis is a pathology that preferentially affects women, with a multifactorial etiology, thus, carrying out a more detailed study of the combination of therapies can be beneficial for the development of a more efficient treatment protocol, ensuring more satisfactory aesthetic results.
4. MATERIALS AND METHODS

   The participants, after selection, will be guided about the procedures to be performed and will sign the Free and Informed Consent Term (TCLE). They were then submitted to assessment using the PAFEG, validated by Meyer et al. (2005), which is a data collection instrument that allows evaluating the degree of cellulite and the levels of sensory alterations resulting from this condition, and later, the

   CELLUQOL summary questionnaire, validated by Hexsel et al. (2011), to assess the quality of life of volunteers.

   The registration of photos will be carried out in orthostatism and in posterior and lateral views (right and left). The camera used will be the same in all the photos and will be positioned on a tripod at a height of 66 cm from the floor, it will be placed at a distance of 55 cm from the volunteer, for better visualization and standardization of the photos. In the same position, photography with a thermographic camera will be carried out.

   Subsequently, they will undergo an ultrasound examination of the affected region. The exam will be carried out with the volunteers positioned in the prone position, in the gluteal and posterior region of the thigh, in an area of 10 cm², which will be delimited by a mold made of rubber E.V.A. A high-frequency ultrasound device (12MHZ) model XG, Samsung brand will be used. The volunteers will also undergo an evaluation of magnetic resonance, which will investigate changes related to cellulite in the skin's architecture, as described in previous studies.
5. PROCEDURES

   For the treatment, the volunteers will receive 15 sessions in total, being held 3 times a week, lasting 50 minutes. The treatment protocol was distributed as follows:

   Session 1 - Manual therapy only Sessions 2 to 6 - Carboxytherapy and phototherapy or radiofrequency Session 7 - Manual therapy only Sessions 8 to 14 - Carboxytherapy and phototherapy or radiofrequency Session 15 - Manual therapy only

   Volunteers will be instructed to wear compressive shorts during treatment. The interventions will be performed using Ibramed™ Carboxitherapy equipment, model Aires™, phototherapy equipment from Ibramed™, model Antares™, radiofrequency equipment from Ibramed™, model Neartek™ In the end, the volunteers will answer the adapted questionnaires from the analysis of patient satisfaction, Segot-chicq et al. (2007) and the Global Aesthetic Improvement Scale - GAIS, by Narins (2003), which is used to classify the response to treatments, allowing a comparative assessment at different times after the therapeutic intervention. The reassessment will be made after the last session, with the repetition of all the procedures mentioned and photos.

   The volunteers will be seen in a dermatofunctional physical therapy treatment outpatient clinic adequately structured for the proposed study, containing an appropriate environmental refrigeration system and good hygiene and lighting conditions, in accordance with the standards of the local Health Surveillance, it will be at the physical therapy clinic, located at Av. Antônio Basílio - Lagoa Seca/ Natal-RN owned by Dr. Eneida Carreiro.
6. DATA ANALYSIS

The collected data will be organized in Excel tables, quantitative data will be submitted to statistical analysis. Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS) version 17.0 for Windows. First, the Kolmogorov-Smirnov(K-S) test was performed to verify the normality of the data. In inferential statistics, the Two-way ANOVA variance test with repeated measures will be used to verify differences between the groups before and after the interventions. Throughout the statistical analysis, a significance level of 5% and a confidence interval of 95% (95% CI) will be assigned. Qualitative data (descriptive analysis of ultrasound and magnetic resonance images) will be described based on medical reports.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* aged between 35 and 55 years old
* multiparous or nulliparous
* using or not contraceptives
* sedentary.

Exclusion Criteria:

* sensitivity disorder during treatment
* do not adapt to the research times and procedures
* abnormalities in blood clotting (coagulopathy)
* use anticoagulants
* polyneuropathies
* pregnant women
* primary malignant disease (tumors) in the treatment area.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Degree of cellulite | 5 weeks post intervention
  Grade of skin lumpiness or skin surface dimpling often seen on the thighs, buttocks and abdomen. It is due to protrusion of subcutaneus fat into the dermis layer of skin.
Levels of sensory alterations | 5 weeks post intervention
  Absent or reduced sensitivity to cutaneous stimulation.

SECONDARY OUTCOMES:
Functionality | 5 weeks post intervention
  Degree of functionality in activities of daily living presented by people with cellulite (assessed with the CELLUQOL questionnaire).The CELLUQOL questionnaire that will be used in this research, published by Hexsel et al (2011) analyzes how much the cellulite affects the participants' quality of life. Between 22 and 44 points, cellulite does not affect quality of life, between 44 and 66 points, cellulite affects quality of life little, between 66 and 88 points, cellulite reasonably affects quality of life, between 88 and 110 points, cellulite greatly affects quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Potiguar, Natal, Lagoa Nova, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Avram MM. Cellulite: a review of its physiology and treatment. J Cosmet Laser Ther. 2004 Dec;6(4):181-5. doi: 10.1080/14764170410003057. PMID 16020201
- [Result] Narins RS, Brandt F, Leyden J, Lorenc ZP, Rubin M, Smith S. A randomized, double-blind, multicenter comparison of the efficacy and tolerability of Restylane versus Zyplast for the correction of nasolabial folds. Dermatol Surg. 2003 Jun;29(6):588-95. doi: 10.1046/j.1524-4725.2003.29150.x. PMID 12786700
- [Result] Rossi AB, Vergnanini AL. Cellulite: a review. J Eur Acad Dermatol Venereol. 2000 Jul;14(4):251-62. doi: 10.1046/j.1468-3083.2000.00016.x. PMID 11204512
- [Result] Segot-Chicq E, Compan-Zaouati D, Wolkenstein P, Consoli S, Rodary C, Delvigne V, Guillou V, Poli F. Development and validation of a questionnaire to evaluate how a cosmetic product for oily skin is able to improve well-being in women. J Eur Acad Dermatol Venereol. 2007 Oct;21(9):1181-6. doi: 10.1111/j.1468-3083.2007.02193.x. PMID 17894702
- [Result] Young VL, DiBernardo BE. Comparison of Cellulite Severity Scales and Imaging Methods. Aesthet Surg J. 2021 May 18;41(6):NP521-NP537. doi: 10.1093/asj/sjaa226. PMID 32785706
- [Result] Zelickson BD, Kist D, Bernstein E, Brown DB, Ksenzenko S, Burns J, Kilmer S, Mehregan D, Pope K. Histological and ultrastructural evaluation of the effects of a radiofrequency-based nonablative dermal remodeling device: a pilot study. Arch Dermatol. 2004 Feb;140(2):204-9. doi: 10.1001/archderm.140.2.204. PMID 14967794
- [Result] Atiyeh BS, Dibo SA. Nonsurgical nonablative treatment of aging skin: radiofrequency technologies between aggressive marketing and evidence-based efficacy. Aesthetic Plast Surg. 2009 May;33(3):283-94. doi: 10.1007/s00266-009-9361-9. Epub 2009 May 13. PMID 19437070
- [Result] Barolet D. Light-emitting diodes (LEDs) in dermatology. Semin Cutan Med Surg. 2008 Dec;27(4):227-38. doi: 10.1016/j.sder.2008.08.003. PMID 19150294